CLINICAL TRIAL: NCT01477307
Title: Effect of Dietary Intervention on Intestinal Microbiota in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Dietary Intervention and Intestinal Microbiota in Non-alcoholic Fatty Liver
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Head, Clinical Nutrition, University Hospital, Geneva
Other Study IDs: 10-231
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: obesity; non-alcoholic fatty liver disease
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hypocaloric diet: The included patients are assigned to a hypocaloric standardized diet for 3 weeks.
  Interventions: Other: Hypocaloric diet

INTERVENTIONS:
Other: Hypocaloric diet — Eurodiet,standardized hypo-caloric diet, during 3 weeks
  Other Names: eurodiet 2

SUMMARY:
In patients with NAFLD/NASH, changes in liver lipid composition and function tests following a short dietary intervention are associated with changes in gut microbiota

DETAILED DESCRIPTION:
Study Hypothesis: In patients with NAFLD/NASH, changes in liver lipid composition and function tests following a short dietary intervention are associated with changes in gut microbiota

Study period:

* Study duration for the participant: 7-10 weeks (1-4 weeks screening period, 3 weeks of intervention + 3 weeks of follow-up)
* Expected study completion date: 30.04.2012 Study type: Single arm before-after study

Number of patients:

20 subjects with obesity and NAFLD / NASH

Main criteria for inclusion:

* Obesity defined as BMI>30
* Abnormal liver function tests defined as ALT > 1.5 times the upper limit of normal
* NAFLD present at liver biopsy
* Age > 18 years, < 60 years

Main exclusion criteria:

* Inability or unwillingness to give consent
* Parenteral nutrition or other ongoing dietary intervention
* Bulimia
* Other known cause of chronic liver disease, including hepatitis B or C, iron overload,
* Use of substances known to alter intestinal permeability, including alcohol and NSAIDs

Intervention:

The phase 2 Eurodiet® program will be used as standardized hypo-caloric diet during a 3-weeks intervention period. The products are commercially available and prescribed to reach 1000 kcal/day. These products will be offered free of charge.

Primary Objective:

To assess the impact of dietary intervention on the relative abundance of fecal Bacteroidetes (expressed as the bacteroidetes to firmicutes ratio) in patients with obesity, abnormal liver function tests and NAFLD

Secondary Objectives:

1. To compare fecal microbiota from patients with NAFLD or NASH at baseline
2. To assess fecal microbiota changes in patients with NAFLD or NASH after dietary intervention
3. To measure liver fat content at baseline and after dietary intervention
4. To assess changes in liver function tests and ultrasensitive CRP, cytokines and serum LPS in relation to changes in microbiota and liver lipid composition
5. To measure orocecal transit time, an index of intestinal pullulation, at baseline and after dietary intervention in patients with NAFLD or NASH
6. To measure intestinal permeability at baseline and after dietary intervention in patients with NAFLD or NASH
7. To assess body composition changes in relation to changes in microbiota and liver lipid composition

Statistical methods:

Baseline and end-of-treatment changes for both bacterial genders and subspecies will be compared using paired-sample Wilcoxon signed-rank test. ANOVA and paired t-test for comparison of other changes within groups. Pearson or Spearman tests will be used to assess correlations between changes in microbiota and changes in liver fat content, liver function tests, CRP, cytokines and intestinal pullulation and permeability.

Sample size:

20 patients with NAFLD/NASH will be studied before and after dietary intervention.

Assessment of end-points:

Fecal microbiota will be analysed with 454-Flex metagenomics Ultrasensitive CRP and serum LPS changes as compared with baseline Serum cytokines as measured with ELISA Liver fat content and composition will be measured using MR spectroscopy Small intestinal overgrowth and intestinal permeability will be assessed using standard 13C breath tests and polyethyleneglycol absorption test Body mass composition changes will be assessed using bioelectrical impedance analysis

Safety :

All adverse events will be recorded throughout the study, in compliance with GCP ICH E6 and national regulations.

ELIGIBILITY:
Inclusion Criteria:

Obesity defined as BMI>30 Abnormal liver function tests defined as ALT > 1.5 times the upper limit of normal NAFLD present at liver biopsy Age > 18 years, < 60 years

Exclusion Criteria:

Inability or unwillingness to give consent Bulimia Other known cause of chronic liver disease, including hepatitis B or C, iron overload, Use of substances known to alter intestinal permeability, including alcohol and NSAIDs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obesity defined as BMI>30 Abnormal liver function tests defined as ALT > 1.5 times the upper limit of normal NAFLD present at liver biopsy Age > 18 years, < 60 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
abundance of fecal abundance of fecal Bacteroidetes | thrice, at inclusion, day 21 and day 42
  Bacterial cells/g caecal content

SECONDARY OUTCOMES:
liver fat content | twice, at inclusion and day 21
  picsel/uni MRI
liver function tests | four times, at screening, inclusion, day 21 and day 42
  mmol/l
CRP | thrice, at screening, inclusion and day 21
  mg/l
serum cytokines | twice, at inclusion and day 21
  ng/ml
serum LPS | twice, at inclusion and day 21
  pg/ml
Breath test pullulation | twice, at inclusion and day 21
intestinal permeability | twice, at inclusion and day 21
  Polyethylene glycol 3350/Polyethylene glycol 400 ratio
body composition | thrice, at inclusion, day 21 and day 42
  body composition in kg and % of body weight
liver lipid composition (biopsy) | once, at screening

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Pataky Z, Genton L, Spahr L, Lazarevic V, Terraz S, Gaia N, Rubbia-Brandt L, Golay A, Schrenzel J, Pichard C. Impact of Hypocaloric Hyperproteic Diet on Gut Microbiota in Overweight or Obese Patients with Nonalcoholic Fatty Liver Disease: A Pilot Study. Dig Dis Sci. 2016 Sep;61(9):2721-31. doi: 10.1007/s10620-016-4179-1. Epub 2016 May 3. PMID 27142672
- See also: Geneva university hospital — http://www.hug-ge.ch/